CLINICAL TRIAL: NCT01332162
Title: CArdiac Desynchronization In Obstructive Hypertrophic CardioMyopathy
Brief Title: CArdiac Desynchronization In Obstructive HCM, CARDIO-HCM
Acronym: CARDIO-HCM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Brugada, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRT-01-2011-HCPB
Record Dates: First submitted 2011-04-01; First posted 2011-04-08 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy (HOCM)
Keywords: Hypertrophic Obstructive Cardiomyopathy (HOCM); Pacing
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biventricular pacing (Experimental): All patients will be pacing during two years
  Interventions: Device: Biventricular pacing
- No Pacing during the first year (Active Comparator): No Pacing during the first year. In the second year all patients will be pacing
  Interventions: Device: No Pacing

INTERVENTIONS:
Device: Biventricular pacing — All patients will be pacing during two years
  Other Names: CRT-D and CRT-P devices:; Promote Quadra CD3239-40, CD3239-40Q. St. Jude Medical; Promote Q CD3221-36. St. Jude Medical; Pacemaquer:; Anthem PM3112. St. Jude Medical
  Arms: Biventricular pacing
Device: No Pacing — No Pacing during the first year. In the second year all patients will be pacing
  Other Names: CRT-D and CRT-P devices:; Promote Quadra CD3239-40, CD3239-40Q. St. Jude Medical; Promote Q CD3221-36. St. Jude Medical; Pacemaquer:; Anthem PM3112. St. Jude Medical
  Arms: No Pacing during the first year

SUMMARY:
The purpose of this study is to evaluate the benefit of the optimal pacing configuration, including the possibility of biventricular or left ventricular pacing, in hypertrophic obstructive cardiomyopathy patients.

DETAILED DESCRIPTION:
In this study, subjects will be randomized to Cardiac Resynchronization Therapy-Defibrillation (CRT-D) or Cardiac Resynchronization Therapy-Pacing (CRT-P) vs Pacing Therapy AAI. Randomization will be stratified by indication. Optimal pharmacological therapy in both treatment arms. Length of follow-up for each subject will be 2y, since all subjects will be followed to a common study termination date.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertrophic Obstructive Cardiomyopathy with significant left ventricular obstruction (baseline LVOT gradient more 50mmHg and severe symptoms

Exclusion Criteria:

* HOCM intraventricular gradient < 50mmHg
* LV ejection fraction < 50%
* mild symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Left ventricular mass and resting left ventricular outflow tract gradient (mmHg). | 1 and 2 years
  Change from Baseline in Left ventricular mass and resting left ventricular outflow tract gradient (mmHg)

SECONDARY OUTCOMES:
Change from Baseline in Clinical evaluation of NYHA,QoL,6MWT,interventricular septum thickness,posterior wall thickness,provoked left ventricular outflow tract gradient,mitral regurgitation grade. | 1 and 2 years
  Change from Baseline in Clinical evaluation (New York Heart Association(NYHA), Quality of life Questionnaire (QoL), 6 Minutes Walk Test (6MWT)), interventricular septum thickness, posterior wall thickness, provoked left ventricular outflow tract gradient, mitral regurgitation grade.

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP BRUGADA, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; ANTONIO BERRUEZO, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain